CLINICAL TRIAL: NCT02397616
Title: Effects of Position and a Test Meal on Esophago-gastric Junction Morphology and Function Assessed by High-resolution Impedance Manometry (HRM)
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-Nr. 2014-0013
Record Dates: First submitted 2015-03-18; First posted 2015-03-25 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Hiatus Hernia
MeSH Terms: conditions — Hernia, Hiatal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: high resolution esophageal manometry — high resolution esophageal manometry using liquid and solid swallows and a test meal.

SUMMARY:
Retrospective analysis for HRM measurements using liquid swallows and a test meal for the presence of hiatal hernia. The investigators will correlate hernia descriptions with presence of acidic reflux and clinical complaints.

DETAILED DESCRIPTION:
We will retrospectively analyze all patients referred to hour unit for high-resolution esophageal manometry. These patients have been tested using liquid swallows and a test meal. We will analyze the HRM measurements for presence of manometric signs of hiatal hernia and determine predictive factors for hernia presence. We will correlate hernia description versus presence of acid reflux, clinical complaints and HRM measurements.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred to our functional lab for esophageal high-resolution manometry from January 2013 - December 20165
* Lack of documentation of patient preferences against usage of medical data for biomedical research
* Male and female patients ≥18 years of age

Exclusion Criteria:

* Age under 18 years
* Patient's wishes against scientific use of their clinical data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to hour unit for high resolution manometry (patients with dysphagia, reflux or other complaints)
Sampling Method: Non-Probability Sample
Enrollment: 380 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Effects of hernia type (consistent hernia, transient hernia and no hernia, as specified bellow) on reflux symptoms | 1 months

SECONDARY OUTCOMES:
Differences in hernia size between sitting and recumbent position as well as between liquid swallows, free drinking and test meal. | 1 hour
Diagnostic accuracy for hernia diagnosis by HRM for sitting, and recumbent position, free drinking and test meal. | 1 hour
Correlation of pH-impedance measurements (if available) with manometric and clinical data. | 1 hour
Correlation of various measurements describing esophageal motility according to Chicago classification with type of hernia, clinical symptoms and pH-impedance measurements | 1 hour
Correlation of hernia diagnosis and hernia size according to imaging exams (if available: CT scan, fluoroscopy) and endoscopy (if available) with hernia diagnosis by HRM | 1 hour
Correlation of body measurements (body mass index, BMI, waist circumference) of patients with type of hernia, clinical symptoms and pH-impedance measurements | 1 hour
Correlation of visceral sensitivity (determined by balloon inflation) with reflux symptoms | 1 hour
Prediction of reflux symptoms using a model including hernia and esophageal peristalsis characteristics, visceral sensitivity (balloon inflation) and anthropometric measurements | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Gastroenterology, University Hospital Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Ang D, Misselwitz B, Hollenstein M, Knowles K, Wright J, Tucker E, Sweis R, Fox M. Diagnostic yield of high-resolution manometry with a solid test meal for clinically relevant, symptomatic oesophageal motility disorders: serial diagnostic study. Lancet Gastroenterol Hepatol. 2017 Sep;2(9):654-661. doi: 10.1016/S2468-1253(17)30148-6. Epub 2017 Jul 3. PMID 28684262
- [Derived] Hollenstein M, Thwaites P, Butikofer S, Heinrich H, Sauter M, Ulmer I, Pohl D, Ang D, Eberli D, Schwizer W, Fried M, Distler O, Fox M, Misselwitz B. Pharyngeal swallowing and oesophageal motility during a solid meal test: a prospective study in healthy volunteers and patients with major motility disorders. Lancet Gastroenterol Hepatol. 2017 Sep;2(9):644-653. doi: 10.1016/S2468-1253(17)30151-6. Epub 2017 Jul 3. PMID 28684261